CLINICAL TRIAL: NCT04484831
Title: An Acceptance-based Therapy Intervention vs. an Enhanced Care Condition for Weight Loss Among Adolescent Girls With Overweight/Obesity: A Randomized, Controlled Trial
Brief Title: A Trial to Test an Acceptance-based Therapy Program Among Adolescent Girls With Overweight/Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: StayWell (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); WellCare Health Plans, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201701609; K01HL141535 (NIH); PA-16-190 (Other Grant/Funding Number: NIH NHLBI)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Weight Loss; Obesity; Overweight
Keywords: acceptance-based therapy; adolescents; weight; weight loss; obesity; overweight
MeSH Terms: conditions — Weight Loss; Obesity; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABT Weight Loss Intervention (Experimental): Adolescent participants will attend sessions that include nutritional education and physical activity education and build skills in the areas of values clarification, mindfulness, self-regulation skills, acceptance of uncomfortable states, goal-setting, problem solving, and self-monitoring.
  Interventions: Behavioral: ABT Weight Loss Intervention
- Enhanced Care (Placebo Comparator): Adolescent participants will receive handouts on elements of a healthy lifestyle and will participate in a midpoint one-on-one nutrition consultation with a registered dietitian.
  Interventions: Other: Enhanced Care

INTERVENTIONS:
Behavioral: ABT Weight Loss Intervention — This includes 15 sessions that are each 90 minutes in length. Intervention sessions will be weekly for the first 2 months, bi-weekly for the next 2 months, and monthly for the last 2 months.
  Arms: ABT Weight Loss Intervention
Other: Enhanced Care — This includes 15 handouts on elements of a healthy lifestyle and a midpoint one-on-one nutrition consultation with a registered dietitian.
  Arms: Enhanced Care

SUMMARY:
The purpose of this study is to investigate the effects of an acceptance-based therapy weight loss intervention compared with enhanced care for adolescents.

DETAILED DESCRIPTION:
Participants will complete baseline assessments and adolescents will be randomized to either an ABT weight loss intervention or enhanced care.

The intervention will include 15 sessions over 6 months. Enhanced care will include 15 healthy lifestyle handouts over 6 months.

Post-treatment assessments will occur.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between ages 14-19 with overweight or obesity at or above the 85th percentile for sex and age as determined by CDC growth charts

Exclusion Criteria:

* Known pregnancy or plans to become pregnant in the next 2 years
* Plans to move out of the area in the next year
* Autism, any intellectual disability (e.g., down syndrome)
* Any condition prohibiting physical activity
* A diagnosis of cardiovascular disease or diabetes
* Have active cancer or cancer requiring treatment in the past 2 years
* Have active or chronic infections (e.g., HIV or TB)
* Have active kidney disease or lung disease
* An eating disorder or substance abuse disorder
* Having recently begun a course of or changed the dosage of any medications known to affect appetite or body composition
* Weight loss greater than or equal to 5% in the previous 6 months
* If they do not follow the study plan

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle I Cardel, PhD, MS, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 participants completed the informed consent process. 40 continued on to randomization and baseline measurements.
Period: Overall Study
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT Weight Loss Intervention | Enhanced Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Information provided details the mean age of the combined sample, the intervention group, and the control group.
  Years | 15.50 (1.54) | 16.05 (1.54) | 15.78 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  White | 14 | 17 | 31
  Black | 4 | 2 | 6
  Other | 2 | 1 | 3
Highest Parental Education [Count of Participants; unit: Participants]
  Some High School/High School Diploma/GED | 2 | 3 | 5
  Some college/Associate degree | 5 | 4 | 9
  Completed Tech or Vocational School/College Graduate | 3 | 5 | 8
  Graduate or professional degree | 10 | 8 | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.66 (5.53) | 34.68 (7.73) | 33.67 (6.71)

OUTCOME MEASURES:

1. Primary Outcome: BMI Change, 95th BMI Percentile (%)
Description: Changes in weight relative to the BMI at the 95th percentile based on sex-and-age (as a difference in percentage units and/or a difference in BMI units) will be evaluated.
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: Change in the 95th BMI percentile %
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
Number analyzed (Participants) | 19 | 20
Change in the 95th BMI percentile % | -1.11 (5.93) | -0.08 (8.05)

2. Secondary Outcome: Change in Quality of Life
Description: Measurements of quality of life (using the valid Pediatric Quality of Life Inventory assessment: scores 0-100) will be conducted. Higher scores indicate better health-related quality of life.
Time Frame: Baseline; Month 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
Number analyzed (Participants) | 19 | 20
score on a scale | 2.94 (10.86) | 3.12 (11.15)

3. Secondary Outcome: Change in Depression Using the Valid Beck Depression Inventory-II
Description: Depression is measured with the Beck Depression Inventory- II (BDI-II). The BDI-II measures the severity of depression. Each item is assessed on a 4-point ordinal categorical scale (0-3 points) that is specific to the question subject matter being addressed (e.g. sadness, self-criticalness, loss of pleasure, etc), and then answer choices are summed to generate a total score. The BDI-II is reliable and valid in an adolescent population.
  Participants receive a sum-score (ranging from 0-63), which correlates with a certain classification and level of depression. Scores 1-10 (normal ups and downs) and 11-16 (mild mood disturbance) are classified as low. Scores 17-20 (borderline clinical depression) and 21-30 (moderate depression) are classified as moderate. Scores 31-40 (severe depression) and 40+ (extreme depression) are classified as significant.
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
Number analyzed (Participants) | 19 | 20
score on a scale | -2.81 (11.58) | 0.71 (12.26)

4. Secondary Outcome: Change in Anxiety-sensitivity Using the Valid Short Scale Anxiety Sensitivity Index Assessment
Description: Measurements of anxiety-sensitivity (using the valid Short Scale Anxiety Sensitivity Index-3 assessment: scores 0-20) will be conducted. Higher scores indicate higher anxiety-sensitivity.
Time Frame: Baseline; Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
Number analyzed (Participants) | 19 | 20
score on a scale | 1.00 (3.65) | 1.00 (5.63)

ADVERSE EVENTS:
Time Frame: from baseline through study completion (6-months)
Arm/Group | ABT Weight Loss Intervention | Enhanced Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT04484831/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04484831/ICF_001.pdf